CLINICAL TRIAL: NCT07198516
Title: The Improvement Effect of Henggliejin on Fatty Liver in Type 2 Diabetes Patients With Nonalcoholic Fatty Liver: a Multicenter, Prospective, Single Arm Clinical Study
Brief Title: The Improvement Effect of Henggliejin on Fatty Liver in Type 2 Diabetes Patients With Nonalcoholic Fatty Liver:
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024XHYG0020
Record Dates: First submitted 2025-08-17; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: NAFLD; Diabete Type 2
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Add Henggelijing treatment for T2DM patients with NAFLD and oral administration of three or fewer hy (Experimental)
  Interventions: Drug: Addition of Hengge Liejing treatment for 48 weeks

INTERVENTIONS:
Drug: Addition of Hengge Liejing treatment for 48 weeks — Treatment with Hengge Liejing for 48 weeks, drug formulation: tablets. Dosage: 10mg qd, taken orally in the morning, before or after breakfast, for 48 consecutive weeks

SUMMARY:
To evaluate the effect and safety of Henggliejin on fatty liver in type 2 diabetes patients with nonalcoholic fatty liver disease

ELIGIBILITY:
Inclusion Criteria:

* (1) Type 2 diabetes diagnosed according to WHO diagnostic criteria, age ≥ 18 years old, ≤ 70 years old, gender unlimited (2) Diagnosed with NAFLD according to the criteria of the "Guidelines for the Prevention and Treatment of Non alcoholic Fatty Liver Disease (2018 Updated Edition)" (3) Before screening, patients with type 2 diabetes who were treated with single or combined drugs of stable dose (except TZDs, SGLT2i, GLP-1RA, insulin and GKAs) for ≥ 8 weeks and had poor blood glucose control, 7% ≤ HbA1c ≤ 10% (4)BMI≥24 kg/m2 (5) Can understand the content and methods of this study and voluntarily sign an informed consent form

Exclusion Criteria:

* (1) Patients with diabetes other than type 2 diabetes, including type 1 diabetes and gestational diabetes (2) Acute diabetes complications such as diabetes ketosis or ketoacidosis, diabetes hypertonic state, diabetes lactic acidosis or serious chronic diabetes complications (3) Individuals with a history of recurrent urinary tract infections and/or genital infections (as determined by clinical physicians) (4) Alcoholic liver disease (alcohol consumption equivalent to less than 30 g/d for males and less than 20 g/d for females in the past two years) (5) Exclude other liver diseases, such as chronic hepatitis B, chronic hepatitis C, primary cholestatic cirrhosis, ballistic obstructive diseases, drug-induced liver damage, hemochromatosis, hepatolenticular deformation, autoimmune hepatitis (6) Combined cirrhosis, combined liver cancer, HIV positive, drug abuse (7) Drugs (tamoxifen, amiodarone, sodium valproate, methotrexate, glucocorticoid, etc.), total parenteral nutrition, inflammatory bowel disease, celiac disease, hypothyroidism, Cushing's syndrome, β - lipoprotein deficiency, lipoatrophic diabetes, Mauriac syndrome, and other special conditions leading to fatty liver (8) Serious trauma or acute infection that may affect blood glucose control occurred within 4 weeks (9) Individuals who have experienced decompensated heart failure (NYHA grades III and IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, severe arrhythmia, or have undergone cardiac surgery or vascular reconstruction (including coronary artery bypass grafting or percutaneous coronary intervention) within 6 months (10) There are obvious blood system diseases (such as aplastic anemia, myelodysplastic syndrome) or any diseases that cause hemolysis or red blood cell instability (such as malaria, hemolytic anemia) (11) Individuals with severe chronic gastrointestinal diseases, or those who have received treatment that may affect drug absorption (such as gastrointestinal surgery) (12) Uncontrolled hyperthyroidism (13) Individuals with mental or neurological disorders who are unwilling to communicate or unable to fully understand and collaborate (14) Pregnant or lactating women (15) There are any laboratory test indicators that meet the following standards:

  1. Alanine aminotransferase>2.0 times ULN and/or aspartate aminotransferase>2.0 times ULN and/or total bilirubin>2.0 times ULN
  2. Blood ketones>ULN
  3. eGFR <30ml/min/1.73 m2； Note: The formula for calculating eGFR is CKD-EPI (which can be calculated within the WeChat mini program)
  4. Blood creatine kinase>3 times ULN (16) In addition to the above, the researchers have determined that patients who are not suitable to participate in this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
After 48 weeks of Henggeleijing treatment, FIB-4 index values | From enrollment to the end of treatment at 48 weeks

SECONDARY OUTCOMES:
Four indicators of liver fibrosis after 48 weeks of Henggelijing treatment | From enrollment to the end of treatment at 48 weeks"
  FIB-4 index is a non-invasive liver fibrosis assessment tool based on blood indicators and age, mainly used to evaluate the risk of liver fibrosis progression in patients with chronic liver disease. Calculation formula: FIB-4=(age x AST)/(platelet count x √ ALT). When calculating, please note that the units of AST and ALT should be U/L, and the unit of platelet count should be 10 ^ 9/L。 When FIB-4<1.3, it indicates no significant liver fibrosis When 1.3 ≤ FIB-4 ≤ 3.25, there may be moderate liver fibrosis When FIB-4>3.25, there is a high suspicion of advanced liver fibrosis or cirrhosis
Improvement rate of FIB-4 index (FIB-4 index improvement defined as a decrease of ≥ 10% from baseline) after 48 weeks of treatment with Henggeleijing | From enrollment to the end of treatment at 48 weeks"
Changes in visceral fat content compared to baseline after 48 weeks of treatment with Henggelijing | From enrollment to the end of treatment at 48 weeks
  Using DUAL bioimpedance method to identify adipose tissue and subcutaneous fat, and safely and conveniently calculate visceral fat area
The results of glycated hemoglobin after 12, 24, and 48 weeks of Henggeleijing treatment | From enrollment to the end of treatment at 48 weeks
The proportion of HbA1c<7% and HbA1c<6.5% after 12, 24, and 48 weeks of treatment with Henggeleijing | From enrollment to the end of treatment at 48 weeks
Changes in fasting plasma glucose levels compared to baseline after 12, 24, 36, and 48 weeks of treatment with Henggeleijing | From enrollment to the end of treatment at 48 weeks
After 12, 24, 36, and 48 weeks of treatment with Henggeleijing, changes in liver enzyme indicators (including AST, ALT, GGT) compared to baseline were observed | From enrollment to the end of treatment at 48 weeks
After 48 weeks of Henggeleijing treatment, the fat content of the endocardial fat pad | From enrollment to the end of treatment at 48 weeks
  Cardiac ultrasound detection of fat content in endocardial fat pad
Changes in C-peptide levels compared to baseline after 12, 24, and 48 weeks of treatment with Henggelijing | From enrollment to the end of treatment at 48 weeks
Changes in fasting insulin levels compared to baseline after 12, 24, and 48 weeks of treatment with Henggelijing | From enrollment to the end of treatment at 48 weeks
Changes in HOMA-IR index compared to baseline after 12, 24, and 48 weeks of treatment with Henggeleijing | From enrollment to the end of treatment at 48 weeks
Changes in fasting body weight compared to baseline after 12, 24, 36, and 48 weeks of treatment with Henggeleijing | From enrollment to the end of treatment at 48 weeks
Blood pressure changes compared to baseline after 12, 24, 36, and 48 weeks of treatment with Henggeleijing | From enrollment to the end of treatment at 48 weeks
Changes in blood lipid profile (including LDL-C, TG, HDL, TC) compared to baseline after 12, 24, 36, and 48 weeks of treatment with Henggeleijing | From enrollment to the end of treatment at 48 weeks
FIB-4 index after 12,and 24 weeks of Henggeleijing treatment | From enrollment to the end of treatment at 24 weeks

OTHER OUTCOMES:
Incidence of Adverse events checklist(Safety during Henggeleijing treatment) | From enrollment to 14 days after the last administration
  Fill in the adverse event record form truthfully, recording the subjects, follow-up time, coding language, occurrence time, severity, duration, relationship with treatment, measures taken, and outcome of the adverse event